CLINICAL TRIAL: NCT05159128
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of JNJ-75105186 in Healthy Japanese Participants and a Single Dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of JNJ-75105186 in Healthy Chinese Participants
Brief Title: A Study of JNJ-75105186 in Healthy Japanese and Chinese Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR109107; 75105186CRD1001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2021-12-06; First posted 2021-12-15 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Single Ascending Dose (SAD) Cohorts (Experimental): Healthy Japanese participants will receive JNJ-75105186 or matching placebo orally in Cohorts 1-3.
  Interventions: Drug: JNJ-75105186; Other: Placebo
- Part 2: Single Dose (SD) Cohort (Experimental): Healthy Chinese participants will receive JNJ-75105186 or matching placebo orally in Cohort 4.
  Interventions: Drug: JNJ-75105186; Other: Placebo

INTERVENTIONS:
Drug: JNJ-75105186 — JNJ-75105186 will be administered orally in Part 1 and 2.
Other: Placebo — Matching placebo to JNJ-75105186 will be administered orally in Parts 1 and 2.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of JNJ-75105186 after single ascending oral dose administration in healthy Japanese participants and after single oral dose administration in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. If there are abnormalities, they must be consistent with the underlying illness in the study population. This determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel including liver enzymes, other specific tests, blood coagulation, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Body weight not less than 50 kilograms (kg) and body mass index within the range 18 to 30 kg per meter square (kg/m^2) (inclusive)
* A woman must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for at least 90 days after receiving the administration of study intervention
* Must sign an informed consent form (ICF) indicating they understand the purpose of, and procedures required for, the study and is willing to participate in the study
* It is recommended that participants are up to date on age-appropriate vaccinations prior to screening as per routine local medical guidelines. For study participants who received locally-approved (and including emergency use-authorized) Coronavirus Disease of 2019 (COVID-19) vaccines recently prior to study entry, follow applicable local vaccine labeling, guidelines, and standards of care for participants receiving immune-targeted therapy when determining an appropriate interval between vaccination and study enrollment

Exclusion Criteria:

* Had major surgery, (example, requiring general anesthesia) within 3 months before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study or within 12 weeks after the last dose of study intervention administration
* History of surgical resection of the stomach, small or large intestine (excluding appendectomy, cholecystectomy, or resection of benign polyps)
* History of bleeding associated with procedures such as endoscopy or phlebotomy; or use of medications such as nonsteroidal anti-inflammatory drugs or aspirin within 28 days prior to screening or planned use during the study
* Preplanned surgery or procedures that would interfere with the conduct of the study
* Clinically significant infection within 30 days prior to screening or any serious infection within 6 months prior to screening requiring intravenous antimicrobial therapy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-04-02 (Estimated); Study Completion 2022-04-02 (Estimated)

PRIMARY OUTCOMES:
Part 1 and 2: Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 6 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Part 1 and 2: Plasma Concentration of JNJ-75105186 | Predose up to 48 hours postdose (up to Day 3)
  Plasma samples will be analyzed to determine concentrations of JNJ-75105186 using a validated, specific and sensitive method.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Souseikai Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency